CLINICAL TRIAL: NCT00299936
Title: Comparison of PEG Interferon Alfa-2b Plus Ribavirin Given as a Fixed Dose or on a Weight Optimized Basis for Treatment of Chronic Hepatitis C in Previously Untreated Adult Subjects
Brief Title: Comparison of PEG-Intron and Two Different Doses of Ribavirin for the Treatment of Chronic Hepatitis C In Treatment Naïve Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Schering-Plough (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P02314; WIN-R
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Last update posted 2006-03-07 (Estimated); Status verified 2006-03

CONDITIONS: Chronic Hepatitis C
Keywords: hepatitis C; chronic hepatitis C; ribavirin; WIN-R
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Ribavirin; peginterferon alfa-2b

INTERVENTIONS:
Drug: Ribavirin, PEG-Intron

SUMMARY:
The purpose of this study is to compare PEG-interferon alfa-2b and two different doses of rivavirin for the treatment of chronic hepatitis C in previously untreated adult subjects

DETAILED DESCRIPTION:
Primary Objective:

This study will evaluate the safety and efficacy of two different PEG-interferon and Ribavirin regimens in patients who have not previously been treated for Hepatitis C. Patients have an equal chance to assignment to one of two treatment arms:

Treatment Arm A:

PEG-interferon 1.5 mcg/kg2 QW + Ribavirin 800 mg/day

OR

Treatment Arm B:

PEG-interferon 1.5mcg/kg2 QW + Ribavirin 800 to 1400 mg/day

Arm A & Arm B: Duration of treatment will be 48 weeks for genotype 1 patients and 24 or 48 weeks for genotype 2 or 3 patients.

ELIGIBILITY:
Adult naive subjects with a diagnosis of compensated chronic hepatitis C (HCV RNA+) who have not previously been treated with interferon, PEG-interferon, ribavirin, or combination interferon + ribavirin are being selected for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000

CONTACTS AND LOCATIONS:
Overall Officials: Ira M Jacobson, MD, Principal Investigator — Weill Medical College of Cornell University

REFERENCES:
- [Derived] Hu KQ, Freilich B, Brown RS, Brass C, Jacobson IM. Impact of Hispanic or Asian ethnicity on the treatment outcomes of chronic hepatitis C: results from the WIN-R trial. J Clin Gastroenterol. 2011 Sep;45(8):720-6. doi: 10.1097/MCG.0b013e31820d35e3. PMID 21836471
- [Derived] Jacobson IM, Brown RS Jr, McCone J, Black M, Albert C, Dragutsky MS, Siddiqui FA, Hargrave T, Kwo PY, Lambiase L, Galler GW, Araya V, Freilich B, Harvey J, Griffel LH, Brass CA; WIN-R Study Group. Impact of weight-based ribavirin with peginterferon alfa-2b in African Americans with hepatitis C virus genotype 1. Hepatology. 2007 Oct;46(4):982-90. doi: 10.1002/hep.21670. PMID 17894323
- [Derived] Jacobson IM, Brown RS Jr, Freilich B, Afdhal N, Kwo PY, Santoro J, Becker S, Wakil AE, Pound D, Godofsky E, Strauss R, Bernstein D, Flamm S, Pauly MP, Mukhopadhyay P, Griffel LH, Brass CA; WIN-R Study Group. Peginterferon alfa-2b and weight-based or flat-dose ribavirin in chronic hepatitis C patients: a randomized trial. Hepatology. 2007 Oct;46(4):971-81. doi: 10.1002/hep.21932. PMID 17894303